CLINICAL TRIAL: NCT00097539
Title: Genentech National Cooperative Growth Study (NCGS) Post-Marketing Surveillance Program For Nutropin AQ® (Somatropin [rDNA Origin] Injection), Nutropin® (Somatropin [rDNA Origin] for Injection), and Protropin® (Somatrem for Injection)
Brief Title: National Cooperative Growth Study (NCGS): A Post-marketing Surveillance Program for Nutropin, Nutropin AQ, Nutropin Depot, and Protropin
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85-036; NCT00231361 (obsolete NCT alias); NCT00672126 (obsolete NCT alias)
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Growth Disorders
Keywords: Pediatric growth disorders
MeSH Terms: conditions — Growth Disorders | interventions — somatrem; Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants With Growth Disorders: Participants initiating therapy with Genentech GH products: Protropin (somatrem for injection), Nutropin (somatropin for injection), Nutropin AQ (somatropin for injection), and Nutropin Depot (somatropin for injectable suspension) for the treatment of pediatric growth disorders as determined by their physician and who have consented to participate in the NCGS will be enrolled in the study and will be followed throughout their course of treatment, or until withdrawal from the NCGS.
  Interventions: Biological: Somatrem; Biological: Somatropin

INTERVENTIONS:
Biological: Somatrem
  Other Names: Protropin
Biological: Somatropin
  Other Names: Nutropin®, Nutropin AQ®, Nutropin Depot™

SUMMARY:
The purpose of this multicenter, open-label, observational, post-marketing surveillance study is to collect long term safety and efficacy information on growth hormone (GH) products: Protropin (somatrem for injection), Nutropin (somatropin for injection), Nutropin AQ (somatropin for injection), and Nutropin Depot (somatropin for injectable suspension) in the treatment of pediatric growth disorders for which GH is prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Participants with open epiphyses
* Children of either sex who are treated with Nutropin Depot, Nutropin AQ, Nutropin, or Protropin for the treatment of growth failure
* Participants who are willing to keep follow up appointments throughout the study participation

Exclusion Criteria:

* Participants treated with a non-Genentech GH preparation
* Participants with closed epiphyses
* Participants with active neoplasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants initiating therapy with Genentech GH products for the treatment of pediatric growth disorders as determined by their physician and who have consented to participate in the NCGS will be enrolled in the study and will be followed throughout their course of treatment, or until withdrawal from the NCGS.
Sampling Method: Non-Probability Sample
Enrollment: 65205 (Actual)
Dates: Start 1985-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were assigned to a growth failure etiology group. Assignment was determined from etiology and medical history data and comments from all participant forms. Etiology groups were mutually exclusive. Participants with multiple etiologies were prioritized as follows: Turner, Renal, Other, Organic GHD, IGHD, ISS, and Undefined.
Groups:
- Idiopathic Growth Hormone Deficiency (IGHD): Participants with IGDH who initiated therapy with Growth Hormone (GH) products (somatrem for injection [Protropin], somatropin for injection [Nutropin, Nutropin AQ, and Nutropin Depot]) and who consented to participate in the National Cooperative Growth Study (NCGS) were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. IGDH etiology group included participants with: Documented IGHD (a maximum GH stimulation test result of less than 10 nanograms per milliliter [ng/mL], coupled with a specific diagnosis of IGHD or equivalent condition by the attending physician; Undocumented IGHD (a stimulation test results were not available, but had a physician diagnosis specifically stated as IGHD or equivalent condition in text); or Presumed IGHD (a stimulation result of less than 10 ng/mL, coupled with the absence of any identifiable criterion for assignation to another etiology grouping).
- Organic Growth Hormone Deficiency (GHD): Participants who initiated therapy with GH products and who consented to participate in the NCGS were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. Organic GHD etiology group included participants with conditions that have a direct effect on the ability of the pituitary gland to modulate GH production, including craniopharyngioma, central nervous system (CNS) tumors, CNS trauma, irradiation, septo-optic dysplasia, and effects of treatments given to participants with leukemia. Inclusion was determined by enrollment form etiology and medical history checkboxes coupled with examination of all participants text.
- Idiopathic Short Stature (ISS): Participants with ISS who initiated therapy with GH products and who consented to participate in the NCGS were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. Participants must have had a stimulation result of greater than or equal to (>/=) 10 ng/mL and/or other identifiable relevant medical text related to ISS. Participants without any identifiable criterion for assignation elsewhere, coupled with a stimulation result of >/=10 ng/mL were assigned to this group. ISS participant may have been Documented ISS, Undocumented ISS, or Presumed ISS, based on text criteria and GH stimulation result of >/=10 ng/mL.
- Turner Syndrome: Participants with Turner Syndrome who initiated therapy with GH products and who consented to participate in the NCGS were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. Participants were assigned to this group, based on medical review of selected participants text, karyotype data, and medical history in cooperation with the NCGS medical advisor.
- Renal Disease: Participants who initiated therapy with GH products and who consented to participate in the NCGS were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. Renal etiology group included participants with chronic renal insufficiency (CRI) or End Stage Renal Disease (ESRD) prior to transplantation as indicated by the CRI/ESRD checkbox on the current NCGS enrollment form or Chronic Renal Disease checkbox (RENAL) from older versions. A search for equivalent terminology in the medical text was also done.
- Other Etiology: Participants who initiated therapy with GH products and who consented to participate in the NCGS were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. The other etiology group represents a heterogeneous mix of participants. Classification in this grouping was determined by examination of enrollment form etiology and medical history checkboxes coupled with examination of participant medical text for selected conditions. Participants with a variety of congenital and/or genetic syndromes, such as Noonan syndrome or Prader-Willi syndrome, were largely included in this classification.
- Undefined Etiology: Participants who initiated therapy with GH products and who consented to participate in the NCGS were enrolled and observed. Participants received GH for the treatment of growth failure as determined by their physician. A participants meeting none of the criteria above was classified as Undefined. These included participants with no medically relevant checkbox, no relevant medical text noted on the enrollment or follow-up forms, and no stimulation result available.
Period: Overall Study
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic Growth Hormone Deficiency (GHD) | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Started | 27286 | 9356 | 12519 | 5651 | 2144 | 8010 | 239
Completed | 8220 | 2825 | 3411 | 2066 | 386 | 2118 | 68
Not Completed | 19066 | 6531 | 9108 | 3585 | 1758 | 5892 | 171
Not completed — Status Unknown (Or no final evaluation) | 11959 | 3948 | 5646 | 2170 | 1106 | 3546 | 108
Not completed — Withdrawal by Subject | 925 | 323 | 346 | 217 | 68 | 229 | 3
Not completed — Participant Non-compliant | 2140 | 567 | 1067 | 353 | 136 | 543 | 18
Not completed — Lack of Efficacy | 249 | 122 | 202 | 105 | 45 | 228 | 5
Not completed — Adverse Event | 78 | 133 | 37 | 27 | 30 | 59 | 1
Not completed — Death | 2 | 7 | 0 | 0 | 1 | 3 | 0
Not completed — Reasons Other Than Above | 3602 | 1382 | 1757 | 692 | 361 | 1244 | 34
Not completed — Reason not Specified | 111 | 49 | 53 | 21 | 11 | 40 | 2

BASELINE CHARACTERISTICS:
Population: Safety evaluable population included all participants enrolled in the study.
Groups:
- Idiopathic Growth Hormone Deficiency (IGHD): Participants who meet any one of the following definitions: Documented IGHD; Undocumented IGHD; Presumed IGHD.
- Organic GHD: Participants with conditions that have a direct effect on the ability of the pituitary gland to modulate GH production, including craniopharyngioma, CNS tumors, CNS trauma, irradiation, septo-optic dysplasia, and effects of treatments given to participants with leukemia. Inclusion was determined by enrollment form etiology and medical history checkboxes coupled with examination of all participants text.
- Idiopathic Short Stature (ISS): Participants must have had a stimulation result of >/=10 ng/mL and/or other identifiable relevant medical text related to ISS. Participants without any identifiable criterion for assignation elsewhere, coupled with a stimulation result of >/=10 ng/mL were assigned to this group. ISS participant may have been Documented ISS, Undocumented ISS, or Presumed ISS, based on text criteria and GH stimulation result of >/=10 ng/mL.
- Turner Syndrome: Participants were assigned to this group, based on medical review of selected participants text, karyotype data, and medical history in cooperation with the NCGS medical advisor.
- Renal Disease: Participants with CRI or ESRD prior to transplantation as indicated by the CRI/ESRD checkbox on the current NCGS enrollment form or Chronic Renal Disease checkbox (RENAL) from older versions. A search for equivalent terminology in the medical text was also done.
- Other Etiology: The other group represents a heterogeneous mix of participants. Classification in this grouping was determined by examination of enrollment form etiology and medical history checkboxes coupled with examination of participant medical text for selected conditions. Participants with a variety of congenital and/or genetic syndromes, such as Noonan syndrome or Prader-Willi syndrome, were largely included in this classification.
- Undefined Etiology: A participants meeting none of the criteria above was classified as Undefined. These included participants with no medically relevant checkbox, no relevant medical text noted on the enrollment or follow-up forms, and no stimulation result available.
- Total: Total of all reporting groups
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology | Total
Number analyzed (Participants) | 27286 | 9356 | 12519 | 5651 | 2144 | 8010 | 239 | 65205
Age, Continuous [Median (Full Range); unit: years] — Age was calculated as first GH dose date minus birth date. Minimum ages shown as 0.0 are less than 19 days (0.05 × 365) and have been rounded to tenths. There were some cases when the birth date and the date of first GH dose were the same. Population: Here, 'Number Analyzed' signifies the number of participants with available Age data.
  years
    number analyzed (Participants) | 27278 | 9352 | 12514 | 5651 | 2143 | 8009 | 239 | 65186
    (all) | 11.6 [0.0 to 41.9] | 10.0 [0.0 to 38.6] | 11.8 [0.0 to 24.2] | 10.2 [0.1 to 21.2] | 10.2 [0.0 to 28.8] | 10.1 [0.0 to 37.8] | 10.7 [0.0 to 17.9] | 11.1 [0.0 to 41.9]
Gender [Count of Participants; unit: Participants]
  Female | 6704 | 3426 | 3213 | 5651 | 630 | 3017 | 81 | 22722
  Male | 20582 | 5930 | 9306 | 0 | 1514 | 4993 | 158 | 42483

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died
Time Frame: From October 1985 to June 2010 (overall approximately 24 years and 9 months)
Population: Safety evaluable population
Measure: Number; unit: participants
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Number analyzed (Participants) | 27286 | 9356 | 12519 | 5651 | 2144 | 8010 | 239
participants | 14 | 96 | 4 | 7 | 23 | 38 | 1

2. Primary Outcome: First Year Annualized Growth Rate
Description: Annualized growth rates are expressed as centimeters per year (cm/yr), computed as the change in height (centimeters) divided by the change in age (years). Growth rates were calculated from the date of the first injection (baseline/ enrollment) to the visit closest to 365*1 days after baseline. Visits within 90 days of 365*1 days after baseline may be used. If multiple visits within 90 days were reported then the visit closest to 365*1 days was used. Growth rates less than (<) -1 or greater than (>) 30 cm/yr were excluded. Growth rates from -1 to 0 were set to 0 cm/yr. Growth rates are summarized by etiology group and gender. Only those participants who had non-missing 1-year growth rate data were included in the analysis.
Time Frame: Year 1
Population: Safety evaluable population. Here, 'N' (number of participants analyzed) signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: cm/yr
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Number analyzed (Participants) | 8715 | 3357 | 3910 | 2762 | 715 | 2940 | 73
cm/yr
  Male: number analyzed (Participants) | 6584 | 2140 | 2972 | 0 | 503 | 1911 | 45
  Male | 9.5 (2.7) | 10.3 (4.1) | 8.6 (2.2) |  | 8.9 (3.6) | 9.5 (3.5) | 9.8 (4.3)
  Female: number analyzed (Participants) | 2131 | 1217 | 938 | 2762 | 212 | 1029 | 28
  Female | 9.8 (3.2) | 11.0 (4.8) | 8.7 (2.5) | 8.0 (2.2) | 8.4 (3.4) | 9.4 (3.8) | 9.1 (2.5)

3. Primary Outcome: Second Year Annualized Growth Rate
Description: Annualized growth rates are expressed as cm/yr, computed as the change in height (centimeters) divided by the change in age (years). Growth rates were calculated from the date of the visit closest to 365 days after baseline to the visit closest to 730 days. Visits within 90 days of 365 and 730 days after baseline may be used. If multiple visits within 90 days were reported then the visit closest to 365 or 730 days was used. Growth rates <-1 or >30 cm/yr were excluded. Growth rates from -1 to 0 were set to 0 cm/yr. Growth rates are summarized by etiology group and gender. Only those participants who had non-missing second-year growth rate data were included in the analysis.
Time Frame: Year 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/yr
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Number analyzed (Participants) | 4980 | 2094 | 2090 | 1790 | 371 | 1761 | 40
cm/yr
  Male: number analyzed (Participants) | 3801 | 1342 | 1605 | 0 | 257 | 1148 | 30
  Male | 7.7 (1.8) | 8.0 (2.5) | 7.3 (1.6) |  | 7.2 (2.4) | 7.5 (2.2) | 7.7 (2.4)
  Female: number analyzed (Participants) | 1179 | 752 | 485 | 1790 | 114 | 613 | 10
  Female | 8.0 (2.2) | 8.2 (2.8) | 7.3 (1.7) | 6.6 (1.5) | 7.2 (2.1) | 7.6 (2.4) | 8.0 (2.3)

4. Primary Outcome: Third Year Annualized Growth Rate
Description: Annualized growth rates are expressed as cm/yr, computed as the change in height (centimeters) divided by the change in age (years). Growth rates were calculated from the date of the visit closest to 730 days after baseline to the visit closest to 1095 days. Visits within 90 days of 730 and 1095 days after baseline may be used. If multiple visits within 90 days were reported then the visit closest to 730 or 1095 days was used. Growth rates <-1 or >30 cm/yr were excluded. Growth rates from -1 to 0 were set to 0 cm/yr. Growth rates are summarized by etiology group and gender. Only those participants who had non-missing third-year growth rate data were included in the analysis.
Time Frame: Year 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/yr
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Number analyzed (Participants) | 3314 | 1581 | 1205 | 1290 | 211 | 1210 | 28
cm/yr
  Male: number analyzed (Participants) | 2512 | 998 | 919 | 0 | 148 | 801 | 20
  Male | 7.0 (1.7) | 7.1 (2.2) | 6.6 (1.6) |  | 6.2 (2.4) | 6.8 (1.9) | 6.5 (1.7)
  Female: number analyzed (Participants) | 802 | 583 | 286 | 1290 | 63 | 409 | 8
  Female | 7.1 (1.7) | 7.2 (2.3) | 6.7 (1.7) | 5.9 (1.5) | 6.1 (2.2) | 6.8 (1.9) | 6.3 (2.6)

5. Primary Outcome: Near Adult Height (NAH)
Description: Heights were standardized with height standardized deviation scores (SDS) to enable height comparisons across ages and sexes using methods and height standards found at: http://www.cdc.gov/growthcharts/cdc_charts.htm. NAH were calculated overall and by etiology groups for participants who had both a non-missing value available height z-score and a non-missing enrollment height (EH) SDS, as well as for participants with 3 or more years of GH therapy (GHT ≥3y).
Time Frame: From October 1985 to June 2010 (overall approximately 24 years and 9 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Number analyzed (Participants) | 4828 | 2352 | 1976 | 1940 | 208 | 1494 | 37
SDS
  NAH | -0.9 (1.1) | -1.1 (1.4) | -1.2 (1.0) | -2.0 (1.0) | -2.0 (1.5) | -1.5 (1.3) | -1.3 (1.2)
  EH | -2.5 (1.0) | -2.4 (1.4) | -2.7 (0.8) | -3.1 (0.9) | -3.1 (1.3) | -2.9 (1.4) | -3.0 (1.7)
  NAH GHT ≥3y: number analyzed (Participants) | 3697 | 1764 | 1458 | 1440 | 126 | 1068 | 28
  NAH GHT ≥3y | -0.8 (1.0) | -1.0 (1.4) | -1.1 (1.0) | -1.9 (1.0) | -1.7 (1.4) | -1.5 (1.3) | -1.2 (1.2)
  EH GHT ≥3y: number analyzed (Participants) | 3697 | 1764 | 1458 | 1440 | 126 | 1068 | 28
  EH GHT ≥3y | -2.6 (1.0) | -2.5 (1.4) | -2.7 (0.8) | -3.2 (1.0) | -3.1 (1.2) | -3.0 (1.4) | -3.2 (1.8)

ADVERSE EVENTS:
Time Frame: From October 1985 to June 2010 (overall approximately 24 years and 9 months)
Description: Protocol-mandated adverse events (AEs): all treatment-related AEs, all serious adverse events (SAEs), and all protocol-defined adverse events of special interest (AESIs) were reported.
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) | Organic GHD | Idiopathic Short Stature (ISS) | Turner Syndrome | Renal Disease | Other Etiology | Undefined Etiology
Serious Adverse Events (participants affected / at risk) | 322/27286 | 595/9356 | 100/12519 | 119/5651 | 141/2144 | 255/8010 | 4/239
Other Adverse Events (participants affected / at risk) | 949/27286 | 523/9356 | 385/12519 | 328/5651 | 101/2144 | 357/8010 | 7/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idiopathic Growth Hormone Deficiency (IGHD) (N=27286) | Organic GHD (N=9356) | Idiopathic Short Stature (ISS) (N=12519) | Turner Syndrome (N=5651) | Renal Disease (N=2144) | Other Etiology (N=8010) | Undefined Etiology (N=239)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 1 | 3 | 0 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thymus enlargement (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 5 | 0 | 0 | 0 | 3 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0
Cardiac septal hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 4 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell naevus syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Caudal regression syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cleft palate (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 4 | 0 | 0 | 0
Congenital aplastic anaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
De Lange's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
DiGeorge's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glycogen storage disorder (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gonadal dysgenesis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypochondroplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Low set ears (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
MELAS syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Macrogenia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pectus carinatum (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Retinitis pigmentosa (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Septo-optic dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spina bifida (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spondyloepiphyseal dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Ear canal erythema (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acromegaly (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 7 | 0 | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Precocious puberty (Endocrine disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Testicular failure primary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Virilism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amblyopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 2 | 1 | 1 | 0 | 1 | 2 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Idiopathic orbital inflammation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iris cyst (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Keratoconus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular vascular disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Optic atrophy (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Optic discs blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Panophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papilloedema (Eye disorders) | 10 | 5 | 1 | 6 | 4 | 3 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinopathy proliferative (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 3 | 4 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 1 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 0 | 1 | 4 | 4 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enamel anomaly (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malocclusion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 8 | 1 | 2 | 3 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Short-bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 15 | 29 | 0 | 4 | 5 | 9 | 0
Asthenia (General disorders) | 2 | 2 | 0 | 1 | 1 | 2 | 0
Brain death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calcinosis (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Crepitations (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyst (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 2 | 10 | 0 | 0 | 2 | 9 | 0
Decreased activity (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device failure (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Device malfunction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease recurrence (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0
Drug resistance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 6 | 11 | 0 | 0 | 0 | 4 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 2 | 8 | 0 | 0 | 1 | 3 | 0
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 0
Liquid product physical issue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 7 | 1 | 1 | 2 | 3 | 0
Mass (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
No therapeutic response (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 3 | 1 | 2 | 0
Pain (General disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 1
Peripheral swelling (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Pseudocyst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 12 | 18 | 1 | 1 | 4 | 11 | 0
Sluggishness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Therapeutic response decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Acute graft versus host disease (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Anaphylactoid reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Immune system disorder (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 19 | 0 | 0
Liver transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0
Lung transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 4 | 1 | 3 | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Colostomy infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Disseminated cytomegaloviral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 2 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 3 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 0 | 1 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Herpes simplex pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Infection parasitic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 6 | 0 | 1 | 2 | 2 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 3 | 0 | 0 | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Orchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 5 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 8 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 4 | 16 | 0 | 0 | 2 | 11 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 3 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 7 | 0 | 0 | 4 | 3 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 1 | 0
Shigella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Shunt infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 3 | 0 | 0 | 0 | 3 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 2 | 0
Varicella (Infections and infestations) | 1 | 2 | 1 | 0 | 1 | 1 | 0
Viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 3 | 1 | 1 | 0 | 4 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Complications of bone marrow transplant (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Complications of transplanted liver (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug dose omission (Injury, poisoning and procedural complications) | 6 | 4 | 2 | 0 | 0 | 3 | 0
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 0 | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 2 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metal poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Off label use (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1 | 0 | 3 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1 | 0 | 1 | 0
Ammonia increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Antinuclear antibody positive (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bleeding time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alcohol increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 8 | 1 | 0
Blood electrolytes abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood follicle stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 1 | 0
Blood gonadotrophin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood testosterone increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body height below normal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body temperature decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone density decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 2 | 1 | 1 | 2 | 0 | 1 | 0
Cardiac output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Culture positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Insulin-like growth factor decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insulin-like growth factor increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipids increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Male genital examination abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Red blood cells urine (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid factor (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 7 | 4 | 0 | 1 | 1 | 5 | 0
Weight increased (Investigations) | 5 | 2 | 0 | 1 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 7 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 13 | 2 | 2 | 3 | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 6 | 2 | 3 | 2 | 4 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 2 | 4 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 19 | 0 | 1 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tetany (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 3 | 4 | 1 | 5 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 1 | 3 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 6 | 2 | 1 | 2 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 1 | 1 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0 | 2 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epiphyseal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 17 | 28 | 2 | 7 | 9 | 10 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Growth retardation (Musculoskeletal and connective tissue disorders) | 8 | 3 | 2 | 0 | 2 | 3 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 4 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 0 | 0 | 5 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 1 | 2 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal osteodystrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 22 | 16 | 5 | 14 | 0 | 21 | 0
Sever's disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Winged scapula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 11 | 1 | 0 | 0 | 2 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angiofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 32 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 10 | 2 | 1 | 0 | 2 | 0
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 75 | 0 | 0 | 0 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Erythroleukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7 | 0 | 0 | 0 | 2 | 0
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 1 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 8 | 1 | 0 | 0 | 0 | 0
Glioneuronal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0 | 1 | 0
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8 | 0 | 0 | 0 | 2 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Medulloblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 28 | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 2 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Optic glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 0 | 0 | 0 | 0 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 0 | 1 | 0 | 2 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6 | 0 | 1 | 1 | 0 | 0
Osteosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian dysgerminoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0 | 0 | 0 | 0
Ovarian germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 1 | 0 | 0 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pineal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pinealoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8 | 0 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Primitive neuroectodermal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prolactinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Testicular embryonal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arachnoid cyst (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0
Autism (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign intracranial hypertension (Nervous system disorders) | 11 | 4 | 2 | 4 | 10 | 8 | 1
Benign rolandic epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain mass (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain stem syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system inflammation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 5 | 0 | 0 | 0 | 1 | 0
Clonic convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cranial nerve palsies multiple (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dysstasia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 4 | 5 | 3 | 0 | 0 | 2 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 17 | 32 | 6 | 5 | 6 | 9 | 0
Hemiparesis (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 1
Hyponatraemic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 12 | 3 | 3 | 2 | 2 | 6 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 6 | 0 | 0 | 0 | 2 | 0
Loss of consciousness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Myoclonic epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatic nerve neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 15 | 45 | 4 | 1 | 2 | 11 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinocerebellar disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vasculitis cerebral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 3 | 4 | 2 | 0 | 1 | 3 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 4 | 2 | 0 | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 5 | 2 | 0 | 0 | 3 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hostility (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate affect (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Listless (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Schizophreniform disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staring (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enuresis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 1 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0
Polyuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 7 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Galactocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Testicular atrophy (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 1 | 0 | 4 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 1 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 2 | 5 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0 | 3 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 2 | 4 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 1 | 1 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0 | 1 | 2 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Walking disability (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cleft lip repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limb operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal transplant (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Talipes correction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Aortic dilatation (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 4 | 9 | 4 | 0
Hypotension (Vascular disorders) | 0 | 7 | 0 | 0 | 1 | 2 | 0
Internal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kawasaki's disease (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Superior mesenteric artery syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neurofibromatosis (Congenital, familial and genetic disorders) | 3 | 4 | 0 | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idiopathic Growth Hormone Deficiency (IGHD) (N=27286) | Organic GHD (N=9356) | Idiopathic Short Stature (ISS) (N=12519) | Turner Syndrome (N=5651) | Renal Disease (N=2144) | Other Etiology (N=8010) | Undefined Etiology (N=239)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 9 | 1 | 1 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supravalvular aortic stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 4 | 0 | 2 | 1 | 2 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell naevus syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carpus curvus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clinodactyly (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Congenital anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congenital aplastic anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congenital nail disorder (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysmorphism (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dysplastic naevus syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femoral anteversion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hamartoma (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemihypertrophy (Congenital, familial and genetic disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Micrognathia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Mitochondrial myopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myotonia congenita (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neurofibromatosis (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pectus carinatum (Congenital, familial and genetic disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pterygium colli (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skeletal dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tourette's disorder (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 3 | 3 | 1 | 3 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 3 | 0 | 1 | 0 | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Acromegaly (Endocrine disorders) | 2 | 1 | 0 | 4 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal suppression (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Delayed puberty (Endocrine disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Early menarche (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Growth accelerated (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Growth hormone deficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 9 | 3 | 0 | 2 | 1 | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pituitary cyst (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Precocious puberty (Endocrine disorders) | 2 | 4 | 2 | 0 | 1 | 2 | 0
Testicular failure (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Astigmatism (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Blindness transient (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 4 | 1 | 0 | 1 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dark circles under eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excessive eye blinking (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Eyelid skin dryness (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Night blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular myasthenia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular vascular disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic atrophy (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Optic disc disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Optic discs blurred (Eye disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Panophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papilloedema (Eye disorders) | 5 | 3 | 2 | 1 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 4 | 2 | 0 | 1 | 0 | 0 | 0
Pseudopapilloedema (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Retinal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal pigmentation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 2 | 3 | 0 | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 12 | 5 | 0 | 3 | 2 | 1 | 0
Visual acuity reduced (Eye disorders) | 4 | 5 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 3 | 5 | 0 | 2 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 5 | 6 | 9 | 2 | 7 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 11 | 1 | 4 | 5 | 1 | 4 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 9 | 5 | 3 | 2 | 0 | 3 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 6 | 3 | 7 | 2 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malocclusion (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 16 | 15 | 2 | 6 | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Painful defaecation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth demineralisation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth deposit (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth development disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tooth resorption (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 31 | 18 | 8 | 12 | 3 | 6 | 0
Adverse event (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 7 | 8 | 2 | 2 | 1 | 2 | 0
Calcinosis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 8 | 3 | 3 | 3 | 1 | 1 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Chronic fatigue syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crying (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Decreased activity (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Developmental delay (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Device defective (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device issue (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Drug effect decreased (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Drug ineffective (General disorders) | 14 | 10 | 7 | 15 | 1 | 18 | 1
Drug interaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Drug resistance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Energy increased (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fat tissue increased (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 20 | 20 | 9 | 6 | 1 | 5 | 0
Feeling abnormal (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 4 | 3 | 1 | 0 | 1 | 3 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hunger (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertrophy (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ill-defined disorder (General disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 0
Impaired healing (General disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 5 | 1 | 3 | 1 | 0 | 1 | 0
Injection site atrophy (General disorders) | 11 | 5 | 2 | 2 | 0 | 1 | 0
Injection site bruising (General disorders) | 11 | 3 | 6 | 6 | 1 | 8 | 0
Injection site discolouration (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Injection site discomfort (General disorders) | 4 | 1 | 1 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 7 | 2 | 3 | 3 | 0 | 1 | 1
Injection site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 4 | 0 | 1 | 0 | 1 | 1 | 0
Injection site hypertrophy (General disorders) | 4 | 0 | 3 | 1 | 0 | 1 | 0
Injection site induration (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Injection site mass (General disorders) | 5 | 1 | 2 | 0 | 1 | 0 | 0
Injection site nodule (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 85 | 28 | 33 | 9 | 7 | 21 | 2
Injection site pruritus (General disorders) | 6 | 1 | 1 | 1 | 1 | 0 | 0
Injection site rash (General disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 6 | 0 | 4 | 3 | 0 | 2 | 0
Injection site swelling (General disorders) | 3 | 1 | 2 | 1 | 1 | 0 | 0
Injection site urticaria (General disorders) | 7 | 3 | 5 | 1 | 0 | 4 | 0
Injection site vesicles (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site warmth (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 11 | 11 | 3 | 2 | 2 | 2 | 0
Mass (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Medical device complication (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medical device pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucous membrane disorder (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
No adverse event (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
No therapeutic response (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 2 | 7 | 0 | 6 | 1 | 3 | 0
Oedema peripheral (General disorders) | 7 | 9 | 2 | 11 | 2 | 5 | 0
Pain (General disorders) | 12 | 4 | 4 | 2 | 1 | 6 | 1
Peripheral swelling (General disorders) | 3 | 7 | 2 | 5 | 1 | 3 | 0
Product odour abnormal (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Product quality issue (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 21 | 10 | 4 | 4 | 2 | 10 | 0
Sluggishness (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0
Temperature intolerance (General disorders) | 2 | 3 | 1 | 0 | 0 | 2 | 0
Tenderness (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Therapeutic response decreased (General disorders) | 5 | 1 | 1 | 1 | 0 | 2 | 0
Thirst (General disorders) | 2 | 3 | 2 | 1 | 0 | 0 | 0
Unevaluable event (General disorders) | 0 | 3 | 0 | 1 | 1 | 1 | 0
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 10 | 1 | 2 | 1 | 0 | 3 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Multiple chemical sensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rubber sensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acne pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 1 | 2 | 1 | 0 | 0 | 0
Cat scratch disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 10 | 4 | 1 | 11 | 0 | 4 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 1 | 1 | 0 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 0 | 4 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 4 | 1 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 7 | 1 | 3 | 1 | 0 | 4 | 0
Injection site abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 10 | 5 | 3 | 3 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 4 | 4 | 1 | 8 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 3 | 2 | 2 | 4 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 4 | 3 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 12 | 2 | 3 | 7 | 3 | 4 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 1 | 3 | 6 | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 2 | 2 | 1 | 5 | 0
Varicella (Infections and infestations) | 2 | 3 | 2 | 0 | 0 | 2 | 0
Viral infection (Infections and infestations) | 5 | 4 | 2 | 3 | 0 | 2 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 5 | 2 | 3 | 0 | 2 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug dose omission (Injury, poisoning and procedural complications) | 53 | 9 | 16 | 13 | 2 | 11 | 1
Ear canal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extra dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 0 | 2 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 3 | 1 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Off label use (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Product preparation error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sports injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Underdose (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2 | 0 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0 | 3 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Antibody test positive (Investigations) | 3 | 3 | 0 | 1 | 0 | 0 | 1
Anti-islet cell antibody positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bleeding time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 1 | 1 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 6 | 1 | 0 | 0 | 0 | 1 | 0
Blood corticotrophin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 12 | 0 | 0
Blood follicle stimulating hormone increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 4 | 1 | 0 | 1 | 1 | 0 | 0
Blood gonadotrophin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood luteinising hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood pressure abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 3 | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood prolactin increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 4 | 2 | 1 | 0 | 0 | 1 | 0
Blood urea decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea nitrogen/creatinine ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 2 | 0 | 1 | 2 | 0 | 0 | 0
Body height below normal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bone density decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 6 | 1 | 0 | 5 | 0 | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glucose tolerance test abnormal (Investigations) | 0 | 2 | 1 | 1 | 0 | 0 | 0
Glucose urine (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Insulin-like growth factor decreased (Investigations) | 0 | 7 | 3 | 0 | 0 | 0 | 0
Insulin-like growth factor increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 2 | 0
Intelligence test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipids abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipids increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mean cell haemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mean cell volume decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein urine (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Thyroxine decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Thyroxine free (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Waist circumference increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 14 | 6 | 5 | 4 | 1 | 5 | 0
Weight increased (Investigations) | 12 | 12 | 4 | 4 | 2 | 7 | 0
White blood cell count decreased (Investigations) | 2 | 1 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 3 | 0 | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Body fat disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carbohydrate intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 7 | 7 | 2 | 2 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 0 | 3 | 0
Failure to thrive (Metabolism and nutrition disorders) | 42 | 41 | 41 | 32 | 9 | 40 | 1
Fat intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 6 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 9 | 1 | 2 | 1 | 7 | 0
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 14 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 5 | 2 | 1 | 0 | 0 | 1 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lack of satiety (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Overweight (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 0 | 0 | 2 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0
Underweight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 66 | 32 | 20 | 17 | 3 | 16 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 6 | 6 | 0 | 4 | 0
Bone deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 9 | 5 | 4 | 4 | 1 | 2 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epiphyseal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epiphyses delayed fusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epiphyses premature fusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 5 | 7 | 0 | 3 | 1 | 0 | 0
Epiphysitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 1 | 0 | 0 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Growth retardation (Musculoskeletal and connective tissue disorders) | 30 | 17 | 18 | 9 | 3 | 10 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 4 | 1 | 4 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 3 | 2 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spine flattening (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 2 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 1 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 26 | 5 | 7 | 2 | 1 | 3 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 12 | 11 | 3 | 2 | 5 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prognathism (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 1 | 0 | 0
Renal osteodystrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rib deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 48 | 32 | 25 | 30 | 3 | 30 | 0
Sever's disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone giant cell tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 0 | 0 | 0 | 0 | 0
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medulloblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 7 | 4 | 13 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2 | 1 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Arachnoiditis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Areflexia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Benign intracranial hypertension (Nervous system disorders) | 4 | 3 | 0 | 3 | 1 | 2 | 0
Burning sensation (Nervous system disorders) | 4 | 1 | 0 | 1 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 7 | 3 | 1 | 0 | 0 | 3 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chorea (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Choreoathetosis (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cluster headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 4 | 2 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 15 | 4 | 6 | 3 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 4 | 1 | 1 | 0 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 128 | 72 | 38 | 34 | 8 | 29 | 0
Hemiparesis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 5 | 0 | 0 | 0 | 1 | 0
Judgement impaired (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 5 | 3 | 1 | 0 | 0 | 3 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 12 | 3 | 3 | 3 | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myoclonic epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuromyopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 4 | 3 | 2 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 8 | 1 | 1 | 0 | 0 | 2 | 0
Seizure (Nervous system disorders) | 15 | 23 | 3 | 4 | 0 | 4 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Slow response to stimuli (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Slow speech (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 7 | 2 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Speech disorder developmental (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stupor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 4 | 2 | 2 | 2 | 0 | 0 | 0
Temporal lobe epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 6 | 1 | 0 | 1 | 0 | 2 | 0
Tunnel vision (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 4 | 0 | 0 | 3 | 0 | 2 | 0
Visual field defect (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 6 | 6 | 3 | 2 | 1 | 4 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 5 | 3 | 2 | 2 | 1 | 4 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anticipatory anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 4 | 1 | 1 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asocial behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Compulsions (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 11 | 5 | 3 | 0 | 1 | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysphemia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eating disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encopresis (Psychiatric disorders) | 3 | 1 | 1 | 1 | 0 | 0 | 0
Frustration (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hostility (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypomania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 2 | 1 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 3 | 3 | 2 | 1 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 3 | 1 | 3 | 2 | 2 | 1 | 0
Negativism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Reading disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 4 | 1 | 1 | 1 | 0 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Staring (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tension (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tic (Psychiatric disorders) | 3 | 0 | 2 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 4 | 3 | 3 | 1 | 0 | 4 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glomerulonephritis acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 2 | 2 | 0 | 1 | 2 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 4 | 1 | 0 | 2 | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 5 | 1 | 2 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 7 | 1 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bilateral breast buds (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 3 | 0 | 3 | 0 | 1 | 2 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Enlarged clitoris (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 33 | 7 | 12 | 0 | 0 | 7 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian failure (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Penile swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scrotal erythema (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular disorder (Reproductive system and breast disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 3 | 0 | 3 | 1
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 8 | 4 | 0 | 6 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 1 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0 | 3 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 2 | 0 | 0 | 3 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 2 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 0 | 1 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 13 | 5 | 7 | 0 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 0 | 2 | 0 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 12 | 3 | 8 | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 3 | 0 | 2 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 1 | 1 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotrichosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Koilonychia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 2 | 1 | 4 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 19 | 7 | 9 | 6 | 0 | 5 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 2 | 0 | 3 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 23 | 6 | 6 | 5 | 0 | 2 | 0
Activities of daily living impaired (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Premenarche (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Treatment noncompliance (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suture insertion (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 7 | 2 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vein disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.